CLINICAL TRIAL: NCT04486794
Title: A Clinical Evaluation of the Efficacy and Safety of Hyaluronic Acid (Restylane®) for the Treatment of Tear Trough Deformity
Brief Title: Restylane® for the Treatment of Tear Trough Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-Res-TT
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Tear Trough Eyelid Deformity

STUDY DESIGN:
Intervention Model Description: Patients in this current trial will initially be randomized to either needle or cannula injections, or no treatment (control; ratio 3:3:1, respectively). Subjects will proceed from randomization in parallel assignment. Subjects initially randomized to the control group at Baseline will be randomized to either needle or cannula treatment at Visit 3, Month 1 (crossover). Subjects in the crossover group will then be seen at weeks 2 and 4 post last treatment, as per Schedule 1.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment at baseline (Experimental)
  Interventions: Device: Restylane®
- Treatment at Month 1 (Active Comparator)
  Interventions: Device: Restylane®

INTERVENTIONS:
Device: Restylane® — Hyaluronic acid

SUMMARY:
The aim of this study is to investigate the effectiveness and tolerability of Restylane® for correction of tear trough deformity, using various injection techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Age of 18 years or greater;
3. Indication for treatment of bilateral tear trough deformity;
4. Symmetry of tear trough deformity at baseline;
5. Subjects who understood and signed the Informed Consent Form (ICF) when entering the study, before performing any investigational procedure.

Exclusion Criteria:

1. Prior (<1 year) or planning to undergo any surgery in the corporal area of interest for study;
2. Any type of comorbidity or clinical condition that, at investigator's discretion, could interfere with study assessments;
3. Diabetes mellitus type 1 or type 2;
4. Autoimmune diseases, collagenosis, decompensated endocrine diseases or any disease that, at investigator's discretion, could interfere with study assessments;
5. Using or have used within 3 months drugs such as corticosteroids, immunosuppressants or others collagen-production inhibitors;
6. Initiated use of hormones or change in dose of hormonal replacement therapy within 3 months;
7. Pregnant or breastfeeding, or wishes to get pregnant within the next 12 months, or refuses to use appropriate contraceptive method (in case of women of childbearing potential);
8. Restylane® should not be used in any person who has hypersensitivity to any of the components of the product;
9. Active skin inflammation or infection in or near the treatment area;
10. Possessing any of the contraindications for use of Restylane®;
11. Septal fat herniation;
12. Severe elastosis (e.g., dermatochalasis);
13. Use of Vitamin E, gingko biloba, Aspirin or non-steroidal anti-inflammatory drugs (NSAIDS) within 1 week of treatment.
14. Use of tear trough injections in the last 12 months.
15. Use of anterior midface injections in the last 12 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
GAIS | 1 month
  Improvement via the blinded evaluator-assessed Global Aesthetic Improvement Scale (GAIS), at the one-month follow up visit. Improvement will be considered as any point-increase above 0 (no change).

SECONDARY OUTCOMES:
Adverse events | Baseline to end of study (up to week 10)
  Safety measurements will be evaluated by the incidence, seriousness, severity and relationship with the medical device to adverse events reported, at all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, FRCSC, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No